CLINICAL TRIAL: NCT00473057
Title: Phase I Study of Autologous Bone Marrow Cell Transplantation in Patient With Ischemic Stroke
Brief Title: Study of Autologous Stem Cell Transplantation for Patients With Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); Ministry of Health, Brazil (Other Government); National Research Council, Brazil (Other)
Responsible Party: Charles Andre, MD, PhD, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONEP-10385; CEP-HUCFF/UFRJ-169/03; Proc.-CNPq-55.2201/2005-7
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Infarction, Middle Cerebral Artery
Keywords: acute stroke; middle cerebral artery; autologous transplantation; bone marrow cells; stem cells; cell therapy
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Autologous cell transplantation — Intra-arterial or intravenous delivery of autologous bone marrow cells

SUMMARY:
This is a open label study to assess the safety of autologous bone marrow transplantation in patients with a ischemic stroke in the middle cerebral artery territory within 90 days from symptoms onset.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to evaluate the safety and feasibility of intra-arterial and intravenous injection of autologous bone marrow mononuclear cells in patients in the acute and sub-acute phase (> 3 and < 90 days after symptoms onset) of ischemic cerebral infarct in the middle cerebral artery territory.

Methods: 15 patients with cerebral infarct within the middle cerebral artery territory will be enrolled in this prospective, nonrandomized, open-labeled study. Up to 10 patients will receive up to 500x 10 6 autologous bone marrow cells injected intra-arterially into the middle cerebral artery through percutaneous approach. The procedure is monitored by Transcranial Doppler (TCD) and electroencephalogram (EEG). Other 5 patients will receive up to 500x 10 6 autologous bone marrow cells injected intravenously. Changes in neurological deficits and improvements in functions will be evaluated at baseline and at regular intervals during follow-up ( 4 months). EEG and neuroimaging exams will be performed at baseline and at regular intervals during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ischemic stroke lasting for more than 3 hours and less than 90 days from symptoms onset
* neuroimages exams showing ischemic cerebral infarct in the middle cerebral artery territory
* age between 18 and 75 years old
* NIHSS between 4 and 20
* spontaneous re-canalization of the middle cerebral artery documented by TCD or MRI
* signed informed consent

Exclusion Criteria:

* difficult in obtaining vascular access for percutaneous procedures
* vascular impossibility to reach the middle cerebral artery through percutaneous approach
* severe carotid stenosis( >70%, by Doppler) related to the severe stroke
* neurological worsening (>4 points in the NIHSS ) due to edema or intracerebral hemorrhage
* primary hematological disease
* neurodegenerative disorder
* previous stroke with mRS > 2
* intracardiac thrombosis
* auto-imune disorders
* osteopathies that could increase the risk of bone marrow harvesting procedure
* thrombophilias
* liver failure
* chronic renal failure (creatinine > 2mg/ml)
* life support dependence
* lacunar stroke
* pregnancy
* history of neoplasia or other comorbidity that could impact patient's short-term survival
* any condition that in the judgment of the investigator would place the patient under undue risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Absence of new neurological deficits during the procedure and/or in the 4 months follow-up. | 4 months

SECONDARY OUTCOMES:
Improvement of neurological deficits | 4 months
Improvement in the neuroimaging exams | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles André, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; Gabriel R de Freitas, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; Rosalia Mendez-Otero, Md, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; Lea Mirian Barbosa da Fonseca, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Clementino Fraga Filho/UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil